CLINICAL TRIAL: NCT02781597
Title: Efficacy of Tranexamic Acid in Controlling Hemoptysis, A Randomized Control Trial
Brief Title: Efficacy of Tranexamic Acid in Hemoptysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Balaji Laxminarayanshetty Bellam, junior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEMOP-TXA 23
Record Dates: First submitted 2016-04-17; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Hemoptysis
Keywords: Hemoptysis; Tranexamic acid; VAS score
MeSH Terms: conditions — Hemoptysis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): All patients will receive basic resuscitative measures and standard treatment like assessment and management of Airway, breathing, circulation, antitussives, and blood products. Patients in group T will receive Inj Tranexamic acid in a loading dose of 1 g over 10 min followed by an infusion of 1 g over 8 h.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): All patients will receive basic resuscitative measures and standard treatment like assessment and management of Airway, breathing, circulation, antitussives, and blood products. Patients will receive 0.9% normal saline instead of Tranexamic acid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Patients will receive Inj Tranexamic acid, in IV in a loading dose of 1 g over 10 min followed by an infusion of 1 g over 8 h in 500ml normal saline
  Other Names: TA
  Arms: Tranexamic acid
Drug: Placebo — Patients will receive 0.9% normal saline
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
The purpose of study is to evaluate the efficacy of tranexamic acid in controlling bleeding in patients of hemoptysis and also to evaluate the safety of tranexamic acid.

DETAILED DESCRIPTION:
Hemoptysis is a common problem in India due to high incidence of tuberculosis and also due to post tubercular sequale. Hemoptysis is usually managed conservatively in mild to moderate cases and cases of massive hemoptysis are managed with more definitive treatment options like vessel embolization (bronchial/pulmonary artery) and surgery as a last option. Tranexamic acid is a antifibrinolytic used in many surgeries and trauma patients to control bleeding and it has been shown effective and safe. The purpose of the study is to evaluate the efficacy of tranexamic acid in patients with hemoptysis in controlling bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ongoing hemoptysis
2. Age: 18 years and above

Exclusion Criteria:

1. Pregnant females
2. Females on oral contraceptives
3. Patients on antifibrinolytics
4. Patients with known drug allergy
5. Patients with renal failure
6. Patients requiring intubation during study period
7. Patients with Massive hemoptysis (>600 ml/24 hrs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in severity of hemoptysis | day1 and day2
  Frequency, amount, VAS score Objective assessment using VAS score at admission and at 48 hours.

SECONDARY OUTCOMES:
Intervention needed | 2 days
  Whether intervention needed to control hemoptysis, in the form of bronchial/pulmonary artery embolization or surgery.(Yes/No)
Blood transfusion needed | 2 days
  Number of blood transfused
Hospital stay | Through study completion, an average of 1 year
  Number of days of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Post graduate institute of medical education and research, Chandigarh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: No
Not required at present